CLINICAL TRIAL: NCT04024228
Title: Immunogenicity and Safety of a High-Dose Quadrivalent Influenza Vaccine Administered by the Intramuscular Route in Subjects 60 Years of Age and Older
Brief Title: Study to Assess the Immune Response and the Safety Profile of a High-Dose Quadrivalent Influenza Vaccine (QIV-HD) Compared to a Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) in Europeans Adults 60 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QHD00011; 2019-000655-14 (EudraCT Number); U1111-1225-0952 (Other: UTN)
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Hemagglutinins; Neuraminidase; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Participants randomized in each group were stratified by age (60 to 64 years of age; 65 years of age and older).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participant and the Investigators remained unaware of the treatment assignments throughout the study. An unblinded qualified trial staff member administered the appropriate vaccine but were not involved in the immunogenicity and safety evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: QIV-HD (Experimental): Participants received a single injection of 0.7 milliliters (mL) QIV-HD, intramuscularly (IM) at Day 0.
  Interventions: Biological: High-Dose Influenza Vaccine (split virion, inactivated), Quadrivalent (QIV-HD) 2019-2020 Northern Hemisphere formulation
- Group 2: QIV-SD (Active Comparator): Participants received a single injection of 0.5 mL QIV-SD, IM at Day 0.
  Interventions: Biological: Standard-Dose influenza virus surface antigens (haemagglutinin and neuraminidase), Inactivated, Influenza Vaccine Quadrivalent, 2019-2020 Northern Hemisphere Strains (QIV-SD)

INTERVENTIONS:
Biological: Standard-Dose influenza virus surface antigens (haemagglutinin and neuraminidase), Inactivated, Influenza Vaccine Quadrivalent, 2019-2020 Northern Hemisphere Strains (QIV-SD) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Other Names: Influvac™ Tetra
  Arms: Group 2: QIV-SD
Biological: High-Dose Influenza Vaccine (split virion, inactivated), Quadrivalent (QIV-HD) 2019-2020 Northern Hemisphere formulation — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Arms: Group 1: QIV-HD

SUMMARY:
Primary Objective:

To demonstrate that high-dose quadrivalent influenza vaccine (QIV-HD) induces an immune response that is superior to the responses induced by standard-dose quadrivalent influenza vaccine (QIV-SD) for all 4 virus strains 28 days post-vaccination in participants 60 to 64 years of age and in participants 65 years of age and older.

Secondary Objective:

* Immunogenicity: To further describe the immune response induced by QIV-HD and QIV-SD in all participants by age group, in pooled age groups, and by vaccine group (QIV-HD; QIV-SD).
* Safety: To describe the safety profile of all participants by age group, in pooled age groups, and by vaccine group (QIV-HD; QIV-SD).

DETAILED DESCRIPTION:
Study duration per participant was approximately 6 months including: 1 day of screening and vaccination, an end of study visit and safety follow-up telephone call approximately at Day 28 and Day 180 after vaccination, respectively.

ELIGIBILITY:
Inclusion criteria :

* Sixty years of age and older on the day of inclusion.
* Able to attend all scheduled visits and complied with all trial procedures.

Exclusion criteria:

* Participant was pregnant, or lactating, or of childbearing potential and did not used an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 4 weeks [28 days] preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 02.
* Previous vaccination against influenza (in the previous 6 months) with either the trial vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on Investigator's judgement.
* Alcohol or substance abuse that, in the opinion of the Investigator might interfere with the trial conduct or completion.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature greater than or equal to (>=) 38.0 degree Celsius) on the day of vaccination. A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Personal or family history of Guillain Barré syndrome.
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that was stable at the time of vaccination in the absence of therapy and participants who had a history of neoplastic disease and had been disease free for >= 5 years)

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1539 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (17):
- Belgium (2):
  - Investigational Site Number 0560001, Ghent
  - Investigational Site Number 0560002, Wilrijk
- France (3):
  - Investigational Site Number 2500001, Gières
  - Investigational Site Number 2500004, Paris
  - Investigational Site Number 2500003, Pierre-Bénite
- Germany (5):
  - Investigational Site Number 2760003, Berlin
  - Investigational Site Number 2760005, Berlin
  - Investigational Site Number 2760004, Berlin
  - Investigational Site Number 2760001, Essen
  - Investigational Site Number 2760002, Oldenburg in Holstein
- Italy (2):
  - Investigational Site Number 3800001, Genova
  - Investigational Site Number 3800003, Palermo
- Investigational Site Number 5280001, Utrecht, Netherlands
- Poland (4):
  - Investigational Site Number 6160001, Dębica
  - Investigational Site Number 6160003, Siemianowice Śląskie
  - Investigational Site Number 6160002, Wola
  - Investigational Site Number 6160004, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: QHD00011 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25339&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 active centers in 6 countries. A total of 1539 participants were enrolled and randomized between 28 October 2019 to 15 November 2019.
Pre-assignment Details: A total of 1533 participants were vaccinated in the study.
Groups:
- Group 1: QIV-HD: Participants received a single injection of 0.7 milliliters (mL) high dose quadrivalent influenza vaccine (QIV-HD), intramuscularly (IM) at Day 0.
- Group 2: QIV-SD: Participants received a single injection of 0.5 mL standard-dose quadrivalent influenza vaccine (QIV-SD), IM at Day 0.
Period: Overall Study
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Started (Randomized) | 774 | 765
Vaccinated | 772 | 761
Full Analysis Set (FAS) (FAS included all randomized participants who received the study vaccine and had a post-vaccination blood sample.) | 769 (377 participants (60-64 years) and 392 participants (>=65 years).) | 758 (377 participants (60-64 years) and 381 participants (>=65 years).)
Completed | 770 | 759
Not Completed | 4 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Deviation | 0 | 2
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: QIV-HD: Participants received a single injection of 0.7 mL QIV-HD, IM at Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD | Total
Number analyzed (Participants) | 774 | 765 | 1539
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 379 | 381 | 760
  >=65 years | 395 | 384 | 779
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (5.82) | 66.6 (6.11) | 66.6 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 390 | 775
  Male | 389 | 375 | 764
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 2 | 2 | 4
  White | 758 | 756 | 1514
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Antibodies in Participants Aged 60-64 Years and Greater Than or Equal to (>=) 65 Years
Description: GMTs of anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage).Titers were expressed in terms of 1/dilution.
Time Frame: Day 28 post-vaccination
Population: Analysis was performed on FAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
titers
  A/H1N1: Day 28: 60-64 years: number analyzed (Participants) | 377 | 377
  A/H1N1: Day 28: 60-64 years | 471 [416 to 533] | 248 [217 to 283]
  A/H3N2: Day 28: 60-64 years: number analyzed (Participants) | 376 | 377
  A/H3N2: Day 28: 60-64 years | 303 [262 to 350] | 178 [154 to 206]
  B1: Day 28: 60-64 years: number analyzed (Participants) | 377 | 377
  B1: Day 28: 60-64 years | 497 [450 to 548] | 330 [297 to 367]
  B2: Day 28: 60-64 years: number analyzed (Participants) | 377 | 377
  B2: Day 28: 60-64 years | 766 [690 to 849] | 433 [391 to 480]
  A/H1N1: Day 28: >= 65 years: number analyzed (Participants) | 392 | 381
  A/H1N1: Day 28: >= 65 years | 286 [250 to 326] | 162 [139 to 190]
  A/H3N2: Day 28: >=65 years: number analyzed (Participants) | 392 | 381
  A/H3N2: Day 28: >=65 years | 324 [281 to 374] | 151 [129 to 176]
  B1: Day 28: >=65 years: number analyzed (Participants) | 392 | 381
  B1: Day 28: >=65 years | 405 [366 to 447] | 262 [236 to 291]
  B2: Day 28: >=65 years: number analyzed (Participants) | 392 | 381
  B2: Day 28: >=65 years | 536 [485 to 592] | 305 [274 to 340]
Statistical Analysis 1: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; A/H1N1: 60-64 years; Test type: Superiority — Superiority of GMTs was concluded if the lower limit of the 2-sided 95% Confidence Interval (CI) for the ratio of GMTs was above 1 between groups for each of the comparisons; GMT ratio = 1.90, 95% CI 2-sided [1.58 to 2.28]
Statistical Analysis 2: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; A/H3N2: 60-64 years; Test type: Superiority — Superiority of GMTs was concluded if the lower limit of the 2-sided 95% CI for the ratio of GMTs was above 1 between groups for each of the comparisons; GMT ratio = 1.70, 95% CI 2-sided [1.38 to 2.08]
Statistical Analysis 3: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; B1: 60-64 years; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.51, 95% CI 2-sided [1.30 to 1.74]
Statistical Analysis 4: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; B2: 60-64 years; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.77, 95% CI 2-sided [1.53 to 2.04]
Statistical Analysis 5: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; A/H1N1: >=65 years; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.76, 95% CI 2-sided [1.44 to 2.15]
Statistical Analysis 6: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; A/H3N2: >=65 years; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 2.15, 95% CI 2-sided [1.74 to 2.65]
Statistical Analysis 7: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; B1: >=65 years; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.55, 95% CI 2-sided [1.34 to 1.79]
Statistical Analysis 8: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; B2: >=65 years; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.76, 95% CI 2-sided [1.52 to 2.03]

2. Secondary Outcome: Geometric Mean Titers of Influenza Antibodies Pre-and Post-Vaccination in All Age Group Participants
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage).Titers were expressed in terms of 1/dilution.
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Group 2: QIV-SD: Participants received a single injection of 0.5 mL QIV-SD; IM at Day 0.
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
titers
  A/H1N1: Day 0: number analyzed (Participants) | 768 | 758
  A/H1N1: Day 0 | 48.6 [43.4 to 54.4] | 46.2 [41.4 to 51.7]
  A/H1N1: Day 28 | 365 [333 to 400] | 200 [181 to 222]
  A/H3N2: Day 0: number analyzed (Participants) | 767 | 757
  A/H3N2: Day 0 | 13.3 [12.3 to 14.4] | 13.0 [12.0 to 14.1]
  A/H3N2: Day 28: number analyzed (Participants) | 768 | 758
  A/H3N2: Day 28 | 313 [283 to 347] | 164 [148 to 182]
  B1: Day 0: number analyzed (Participants) | 767 | 757
  B1: Day 0 | 63.9 [57.7 to 70.7] | 74.5 [67.3 to 82.4]
  B1: Day 28 | 447 [417 to 480] | 294 [272 to 316]
  B2: Day 0: number analyzed (Participants) | 765 | 755
  B2: Day 0 | 89.7 [80.5 to 99.9] | 96.6 [86.9 to 107]
  B2: Day 28 | 638 [594 to 686] | 363 [337 to 392]

3. Secondary Outcome: Geometric Mean Titers of Influenza Antibodies Pre- and Post-Vaccination in Participants Aged 60-64 Years and >=65 Years
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Titers were expressed in terms of 1/dilution.
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Group 1: QIV-HD: Participants received a single injection of 0.7 mL QIV-HD; IM at Day 0.
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
titers
  A/H1N1: Day 0: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H1N1: Day 0: 60-64 Years | 50.2 [42.7 to 59.0] | 50.0 [42.6 to 58.8]
  A/H1N1: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  A/H1N1: Day 28: 60-64 Years | 471 [416 to 533] | 248 [217 to 283]
  A/H3N2: Day 0: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H3N2: Day 0: 60-64 Years | 11.5 [10.4 to 12.8] | 12.5 [11.2 to 14.0]
  A/H3N2: Day 28: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H3N2: Day 28: 60-64 Years | 303 [262 to 350] | 178 [154 to 206]
  B1: Day 0: 60-64 Years: number analyzed (Participants) | 377 | 377
  B1: Day 0: 60-64 Years | 54.7 [47.4 to 63.2] | 68.7 [59.4 to 79.5]
  B1: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  B1: Day 28: 60-64 Years | 497 [450 to 548] | 330 [297 to 367]
  B2: Day 0: 60-64 Years: number analyzed (Participants) | 377 | 375
  B2: Day 0: 60-64 Years | 80.4 [68.6 to 94.3] | 93.2 [79.5 to 109]
  B2: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  B2: Day 28: 60-64 Years | 766 [690 to 849] | 433 [391 to 480]
  A/H1N1: Day 0: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H1N1: Day 0: >=65 Years | 47.1 [40.1 to 55.2] | 42.8 [36.6 to 50.0]
  A/H1N1: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H1N1: Day 28: >=65 Years | 286 [250 to 326] | 162 [139 to 190]
  A/H3N2: Day 0: >=65 Years: number analyzed (Participants) | 391 | 380
  A/H3N2: Day 0: >=65 Years | 15.2 [13.5 to 17.1] | 13.5 [12.1 to 15.0]
  A/H3N2: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H3N2: Day 28: >=65 Years | 324 [281 to 374] | 151 [129 to 176]
  B1: Day 0: >=65 Years: number analyzed (Participants) | 390 | 380
  B1: Day 0: >=65 Years | 74.2 [64.3 to 85.6] | 80.7 [70.1 to 92.9]
  B1: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  B1: Day 28: >=65 Years | 405 [366 to 447] | 262 [236 to 291]
  B2: Day 0: >=65 Years: number analyzed (Participants) | 388 | 380
  B2: Day 0: >=65 Years | 99.7 [86.1 to 115] | 100 [86.8 to 115]
  B2: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  B2: Day 28: >=65 Years | 536 [485 to 592] | 305 [274 to 340]

4. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of Influenza Antibodies in All Age Group Participants
Description: GMTRs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). GMTRs were calculated as the ratio of GMTs post-vaccination (on Day 28) and pre-vaccination (on Day 0).
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
ratio
  A/H1N1: Day 28/Day 0: number analyzed (Participants) | 768 | 758
  A/H1N1: Day 28/Day 0 | 7.50 [6.68 to 8.42] | 4.34 [3.88 to 4.84]
  A/H3N2: Day 28/Day 0: number analyzed (Participants) | 767 | 757
  A/H3N2: Day 28/Day 0 | 23.7 [21.4 to 26.1] | 12.6 [11.3 to 14.0]
  B1: Day 28/Day 0: number analyzed (Participants) | 767 | 757
  B1: Day 28/Day 0 | 7.02 [6.34 to 7.77] | 3.95 [3.56 to 4.38]
  B2: Day 28/Day 0: number analyzed (Participants) | 765 | 755
  B2: Day 28/Day 0 | 7.13 [6.44 to 7.90] | 3.77 [3.42 to 4.15]

5. Secondary Outcome: Geometric Mean Titer Ratios of Influenza Antibodies in Participants Aged 60-64 Years and >=65 Years
Description: as for outcome 4
Time Frame: Day 0 (pre-vaccination), Day 28 (post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
ratio
  A/H1N1: Day 28/Day 0: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H1N1: Day 28/Day 0: 60-64 Years | 9.36 [7.86 to 11.1] | 4.96 [4.20 to 5.85]
  A/H3N2: Day 28/Day 0: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H3N2: Day 28/Day 0: 60-64 Years | 26.2 [22.8 to 30.2] | 14.2 [12.2 to 16.6]
  B1: Day 28/Day 0: 60-64 Years: number analyzed (Participants) | 377 | 377
  B1: Day 28/Day 0: 60-64 Years | 9.07 [7.84 to 10.5] | 4.80 [4.11 to 5.60]
  B2: Day 28/Day 0: 60-64 Years: number analyzed (Participants) | 377 | 375
  B2: Day 28/Day 0: 60-64 Years | 9.52 [8.19 to 11.1] | 4.66 [4.03 to 5.39]
  A/H1N1: Day 28/Day 0: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H1N1: Day 28/Day 0: >=65 Years | 6.07 [5.22 to 7.05] | 3.80 [3.27 to 4.41]
  A/H3N2: Day 28/Day 0: >=65 Years: number analyzed (Participants) | 391 | 380
  A/H3N2: Day 28/Day 0: >=65 Years | 21.4 [18.6 to 24.7] | 11.2 [9.66 to 13.0]
  B1: Day 28/Day 0: >=65 Years: number analyzed (Participants) | 390 | 380
  B1: Day 28/Day 0: >=65 Years | 5.48 [4.78 to 6.28] | 3.25 [2.83 to 3.73]
  B2: Day 28/Day 0: >=65 Years: number analyzed (Participants) | 388 | 380
  B2: Day 28/Day 0: >=65 Years | 5.39 [4.72 to 6.15] | 3.06 [2.70 to 3.46]

6. Secondary Outcome: Percentage of Participants (All Age Group Participants) With Neutralizing Antibody Titers >=40 (1/Dilution)
Description: Neutralizing Antibody titer was measured using HAI assay method for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Percentage of participants (all age group participants) with neutralizing antibody titers >=40 (1/dilution) is reported in the outcome measure.
Time Frame: Day 28 post-vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
percentage of participants
  A/H1N1: Day 28 | 96.6 [95.1 to 97.8] | 88.4 [85.9 to 90.6]
  A/H3N2: Day 28: number analyzed (Participants) | 768 | 758
  A/H3N2: Day 28 | 93.8 [91.8 to 95.4] | 86.4 [83.8 to 88.8]
  B1: Day 28 | 99.5 [98.7 to 99.9] | 99.2 [98.3 to 99.7]
  B2: Day 28 | 99.5 [98.7 to 99.9] | 98.3 [97.1 to 99.1]

7. Secondary Outcome: Percentage of Participants (Aged 60-64 Years and >=65 Years) With Neutralizing Antibody Titers >=40 (1/Dilution)
Description: Neutralizing Antibody titer was measured using HAI assay method for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Percentage of participants (aged 60-64 Years and >=65 Years) with neutralizing antibody titers >=40 (1/dilution) is reported in the outcome measure.
Time Frame: Day 28 post-vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
percentage of participants
  A/H1N1: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  A/H1N1: Day 28: 60-64 Years | 98.1 [96.2 to 99.3] | 92.3 [89.1 to 94.8]
  A/H3N2: Day 28: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H3N2: Day 28: 60-64 Years | 94.9 [92.2 to 96.9] | 89.1 [85.5 to 92.1]
  B1: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  B1: Day 28: 60-64 Years | 100 [99.0 to 100] | 99.5 [98.1 to 99.9]
  B2: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  B2: Day 28: 60-64 Years | 99.7 [98.5 to 100] | 99.5 [98.1 to 99.9]
  A/H1N1: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H1N1: Day 28: >=65 Years | 95.2 [92.5 to 97.1] | 84.5 [80.5 to 88.0]
  A/H3N2: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H3N2: Day 28: >=65 Years | 92.6 [89.5 to 95.0] | 83.7 [79.6 to 87.3]
  B1: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  B1: Day 28: >=65 Years | 99.0 [97.4 to 99.7] | 99.0 [97.3 to 99.7]
  B2: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  B2: Day 28: >=65 Years | 99.2 [97.8 to 99.8] | 97.1 [94.9 to 98.6]

8. Secondary Outcome: Percentage of Participants (All Age Group Participants) Achieving Seroconversion Against Antigens
Description: Anti-influenza antibodies were measured by HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Seroconversion was defined as either a pre-vaccination HAI titer less than (<) 1:10 (1/dilution) and a post-vaccination titer >=1:40 (1/dilution) or a pre-vaccination titer >= 1:10 (1/dilution) and a >= four-fold increase in post-vaccination titer at Day 28. Percentage of participants (all age group participants) achieving seroconversion is reported in the outcome measure.
Time Frame: Day 28 post-vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
percentage of participants
  A/H1N1: Day 28: number analyzed (Participants) | 768 | 758
  A/H1N1: Day 28 | 62.1 [58.6 to 65.6] | 39.2 [35.7 to 42.8]
  A/H3N2: Day 28: number analyzed (Participants) | 767 | 757
  A/H3N2: Day 28 | 88.1 [85.6 to 90.3] | 74.2 [71.0 to 77.3]
  B1: Day 28: number analyzed (Participants) | 767 | 757
  B1: Day 28 | 62.5 [58.9 to 65.9] | 41.2 [37.7 to 44.8]
  B2: Day 28: number analyzed (Participants) | 765 | 755
  B2: Day 28 | 62.7 [59.2 to 66.2] | 41.6 [38.0 to 45.2]

9. Secondary Outcome: Percentage of Participants (Aged 60-64 Years and >=65 Years) Achieving Seroconversion Against Antigens
Description: Anti-influenza antibodies were measured by HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B1 (B Victoria lineage), and B2 (B Yamagata lineage). Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 (1/dilution) and a post-vaccination titer >= 1:40 (1/dilution) or a pre-vaccination titer >= 1:10 (1/dilution) and a >= four-fold increase in post-vaccination titer at Day 28. Percentage of participants (aged 60-64 Years and >=65 Years) achieving seroconversion is reported in the outcome measure.
Time Frame: Day 28 post-vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 769 | 758
percentage of participants
  A/H1N1: Day 28: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H1N1: Day 28: 60-64 Years | 66.5 [61.5 to 71.2] | 41.4 [36.4 to 46.5]
  A/H3N2: Day 28: 60-64 Years: number analyzed (Participants) | 376 | 377
  A/H3N2: Day 28: 60-64 Years | 89.4 [85.8 to 92.3] | 76.7 [72.1 to 80.8]
  B1: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 377
  B1: Day 28: 60-64 Years | 68.2 [63.2 to 72.8] | 47.7 [42.6 to 52.9]
  B2: Day 28: 60-64 Years: number analyzed (Participants) | 377 | 375
  B2: Day 28: 60-64 Years | 70.6 [65.7 to 75.1] | 48.5 [43.4 to 53.7]
  A/H1N1: Day 28: >=65 Years: number analyzed (Participants) | 392 | 381
  A/H1N1: Day 28: >=65 Years | 57.9 [52.8 to 62.8] | 37.0 [32.1 to 42.1]
  A/H3N2: Day 28: >=65 Years: number analyzed (Participants) | 391 | 380
  A/H3N2: Day 28: >=65 Years | 87.0 [83.2 to 90.1] | 71.8 [67.0 to 76.3]
  B1: Day 28: >=65 Years: number analyzed (Participants) | 390 | 380
  B1: Day 28: >=65 Years | 56.9 [51.8 to 61.9] | 34.7 [30.0 to 39.8]
  B2: Day 28: >=65 Years: number analyzed (Participants) | 388 | 380
  B2: Day 28: >=65 Years | 55.2 [50.1 to 60.2] | 34.7 [30.0 to 39.8]

10. Secondary Outcome: Number of Participants Reporting Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes post-vaccination
Population: Analysis was performed on safety analysis set (SafAS) which included participants who had received the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 772 | 761
Participants | 2 | 1

11. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the product administered. Solicited injection site reactions included induration, bruising, pain, erythema, and swelling.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on the SafAS population. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 770 | 759
Participants
  Bruising | 12 | 7
  Erythema | 157 | 85
  Induration | 132 | 64
  Pain | 350 | 159
  Swelling | 140 | 62

12. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the product administered. Solicited systemic reactions included fever, headache, malaise, myalgia and shivering.
Time Frame: Within 7 days post-vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 770 | 759
Participants
  Fever | 18 | 4
  Headache | 184 | 141
  Malaise | 164 | 89
  Myalgia | 202 | 93
  Shivering | 128 | 54

13. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Within 28 days post-vaccination
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 772 | 761
Participants | 190 | 172

14. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Including Adverse Event of Special Interest (AESIs)
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. A SAE which caused death of the participant was considered as fatal SAE. Adverse events of special interest (AESIs) was defined as event for which ongoing monitoring and rapid communication by the investigator to the sponsor was done.
Time Frame: From Day 0 up to 6 months post-vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 772 | 761
Participants
  SAE | 17 | 21
  AESI | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected from Day 0 (post-vaccination) up to 28 days post-vaccination. Solicited reaction data were collected up to Day 7 post-vaccination. SAE data were collected throughout the study, i.e. up to 6 months post-vaccination.
Description: Analysis was performed on safety analysis set. A solicited reaction was an adverse reaction that was prelisted (i.e., solicited) in the CRB and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRB in terms of diagnosis and/or onset window post-vaccination. In the AE section, solicited reactions Shivering were reported as Chills.
Groups:
- Group 1 QIV-HD: Participants received a single injection of 0.7 mL QIV-HD, IM at Day 0.
- Group 2 QIV-SD: Participants received a single injection of 0.5 mL QIV-SD, IM at Day 0.
Arm/Group | Group 1 QIV-HD | Group 2 QIV-SD
All-Cause Mortality (participants affected / at risk) | 2/772 | 0/761
Serious Adverse Events (participants affected / at risk) | 17/772 | 21/761
Other Adverse Events (participants affected / at risk) | 507/772 | 354/761
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 QIV-HD (N=772) | Group 2 QIV-SD (N=761)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Gastric Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Corona Virus Infection (Infections and infestations) | 2 (2) | 1 (1)
Pilonidal Cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Vith Nerve Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intermittent Claudication (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 QIV-HD (N=772) | Group 2 QIV-SD (N=761)
Chills (General disorders) | 128 (130) | 57 (58) — Chills/Shivering events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Injection Site Erythema (General disorders) | 157 (158) | 85 (85)
Injection Site Induration (General disorders) | 132 (133) | 64 (64)
Injection Site Pain (General disorders) | 350 (350) | 161 (161) — Pain events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Injection Site Swelling (General disorders) | 140 (140) | 62 (62)
Malaise (General disorders) | 168 (168) | 90 (90) — Malaise events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Myalgia (Musculoskeletal and connective tissue disorders) | 206 (207) | 94 (94) — Myalgia events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Headache (Nervous system disorders) | 190 (196) | 149 (156) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT04024228/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04024228/SAP_001.pdf